CLINICAL TRIAL: NCT02401932
Title: Comparison of Malignant and Non-malignant Disorders Associated Bone Marrow Hemophagocytosis: A Single Center Experience
Brief Title: Retrospective Analysis for Patients With Hemophagocytosis in Bone Marrow
Status: Completed | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2015-02-013
Record Dates: First submitted 2015-03-09; First posted 2015-03-30 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Hemophagocytosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Hemophagocytosis: The group includes patients who have the evidence of hemophagocytosis in their bone marrow or other sites.
  Interventions: Other: Hemophagocytosis

INTERVENTIONS:
Other: Hemophagocytosis — Best supportive care and immunosuppressive treatments

SUMMARY:
Comparison of malignant and non-malignant disorders associated bone marrow hemophagocytosis.

DETAILED DESCRIPTION:
This is a retrospective study comparing malignant and non-malignant disorders associated bone marrow hemophagocytosis. The medical record of patients who had documented evidences of hemophagocytosis in bone marrow are reviewed. The clinical and biological characteristics are compared according to the underlying disorders of hemophagocytosis.

ELIGIBILITY:
Inclusion Criteria:

* patients who had evidence of hemophagocytic histiocytosis in bone marrow aspiration and biopsy

Exclusion Criteria:

* patients who did not evidence of hemophagocytic histiocytosis in bone marrow aspiration and biopsy

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators reviewed the electronic data base of medical records at the Samsung Medical Center, and selected 264 patients who had evidence of hemophagocytic histiocytosis in bone marrow aspiration and biopsy between January 2000 and June 2014.
Sampling Method: Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2014-01; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Overall survival | 12 Months

CONTACTS AND LOCATIONS:
Overall Officials: Seok Jin Kim, MD, PhD, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea